## **COVER PAGE for Statistical Analysis Plan**

Title: Using Pressure Detecting Insoles to Reduce Knee Loading

NCT number: NCT02955225

Document date: May 12, 2015

## Statistical Analysis Plan

To address the primary hypothesis we will use paired t-tests. Separate mixed ANOVAs will be used to evaluate either differences in knee loading or questionnaire scores between the two treatment conditions longitudinally. Pearson or Spearman correlations will be used to evaluate associations between changes in subsections of the KOOS questionnaire and knee loads.